CLINICAL TRIAL: NCT05595629
Title: Implementing an App-based Remote Blood Pressure Monitoring Program to Reduce Health Disparities Among Women With Hypertension During Pregnancy
Brief Title: App-based Remote Blood Pressure Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Adam Lewkowitz, Assistant Professor, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WIH 21-0101
Record Dates: First submitted 2022-10-04; First posted 2022-10-27 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Gestational Hypertension; Preeclampsia; Chronic Hypertension Complicating Pregnancy
Keywords: chronic or gestational hypertension, preeclampsia; remote blood pressure monitoring; smartphone application
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants who consent will be unaware of the existence of the other remote blood pressure monitoring program. The nurse practitioner who manages postpartum hypertension for all participants will be aware of randomization group but will manage each participant per a standard treatment algorithm regardless of randomization group. The research team and outcomes assessors will be blinded to the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-message based remote blood pressure monitoring (Active Comparator): Women in this group will receive current standard of care: remote blood pressure monitoring via text message. Specifically, they will receive automatic blood pressure cuffs, instructions how to obtain their blood pressures and log them into our Electronic Medical Record, and contact information for the nurse practitioner and community health worker managing the program. The NP will respond via text message to each individual measurement with instructions as to next steps.
  Interventions: Behavioral: text-message based remote blood pressure monitoring
- App-based remote blood pressure monitoring (Experimental): Women in this group will receive a Bluetooth-enabled automatic blood pressure cuff that synchs automatically to a smartphone application that incorporates Artificial Intelligence to respond to each recorded measurements with recommended next steps and also document the measurement and response in a secure platform. This affiliated smartphone application will also contain education on hypertension management. Upon receipt of the blood pressure cuff, participants will be instructed to set up the program/app.
  Interventions: Behavioral: App-based remote blood pressure monitoring

INTERVENTIONS:
Behavioral: App-based remote blood pressure monitoring — Fully synched bluetooth-enabled remote blood pressure monitoring using a smartphone application. The digital health company, Twistle, has modified an existing postpartum hypertension pathway in their app according to our hospital's management algorithm.
  Other Names: Twistle
  Arms: App-based remote blood pressure monitoring
Behavioral: text-message based remote blood pressure monitoring — Participants will receive automatic blood pressure cuffs and instructions as to how to upload their measurements to the Electronic Medical Record.
  Arms: Text-message based remote blood pressure monitoring

SUMMARY:
Remote postpartum blood pressure monitoring program with text messages has been shown to increase adherence to recommended postpartum blood pressure checks among those with hypertension at discharge from birth hospitalization, but these programs require medically trained professionals to respond to each individual text message. A bluetooth-enabled blood pressure cuff that synchs automatically a smartphone application that leverages Artificial Intelligence to provide tailored recommendations based on recorded blood pressure measurements--and can also provide on-demand education on hypertension--may be less costly way to provide similar support.

DETAILED DESCRIPTION:
Preeclampsia or gestational hypertension-described as hypertension in pregnancy-affects up to 10% of all pregnancies and is a main driver of maternal morbidity in Rhode Island and the United States. The rates of hypertension in pregnancy have disproportionately affected women of color and may explain why racial minorities have higher maternal morbidity. The American College of Obstetricians and Gynecologists has called for novel interventions to improve health equity and maternal morbidity outcomes among women hypertension in pregnancy. Technology-based interventions (i.e. remote blood pressure monitoring, telehealth visits, text-based communication) have improved access to care but, to date, have not yet demonstrated an effect on reducing maternal morbidity outcomes. It is possible that the lack of effect on maternal morbidity is due to the simplicity of the technology-based interventions previously employed (i.e. text message-based systems). Advanced digital health interventions on blood pressure--namely remote blood pressure monitoring through Bluetooth-enabled blood pressure cuffs and incorporation of a commercially available smartphone application that includes education and patient support as part of a "hypertension in pregnancy pathway"-may more effectively improve perinatal health equity compared to standard SMS-based messaging by reducing perinatal morbidity/mortality among women of color hypertension during their pregnancy.

The investigators propose a pilot randomized control trial to examine the feasibility, acceptability, and preliminary estimates of effects of smartphone application-based (app-based) Bluetooth enabled remote blood pressure monitoring (intervention group) when compared to a SMS (short message system such as text message) based remote blood pressure monitoring group (control group). The investigators' long-term goal is to use the most cost-effective intervention (app-based vs SMS-based remote blood pressure monitoring) to improve health equity and maternal morbidity outcomes for pregnant women with hypertension during pregnancy who live in Rhode Island and beyond. The investigators plan to use pilot data from this proposal to support an efficacy trial powered to detect differences in maternal morbidity outcomes between app-based remote blood pressure monitoring and routine care with SMS monitoring.

In addition, this proposal stems from a hospital-wide effort at Women & Infants Hospital (WIH) to reduce racial disparities among women of color in terms of frequency of severe maternal morbidity (SMM). SMM is a metric created by the Centers for Disease Control and Prevention that includes blood transfusion as well as adverse outcomes ranging from arrhythmia to eclampsia to intubation. SMM associated with hypertension is driven by asymptomatic postpartum hypertension. This is easily identified and managed prior to becoming SMM when patients adhere to recommended blood pressure checks after discharge. Excluding blood transfusion (which does not pertain to hypertension), the overall rate of SMM among women with hypertension during pregnancy who deliver at WIH is 6.6%. However, there is a significant difference along racial and ethnic lines: the rate of SMM in the setting of hypertension among black women is 6.8% compared to 4.5% among white women, and the rate of SMM in the setting of preeclampsia is 9.4% among Hispanic women compared to 4.9% among non-Hispanic women. The overall dual aim of the initiative is to reduce the disparity in rates of SMM among those with hypertension between black and white women and between Hispanic and non-Hispanic women by at least 33% by December 31, 2022. As part of WIH's equity initiative, automatic blood pressure cuffs (non Bluetooth enabled) will be provided to consenting women with hypertension at discharge from delivery hospitalization as part of routine care. In this study, rates of SMM before the hospital-wide implementation of SMS-based remote blood pressure monitoring will be compared to those after. Thus, for this proposal, this proposal exploring whether app-based remote blood pressure monitoring is required to decrease maternal morbidity compared to standard care with remote SMS blood pressure monitoring.

ELIGIBILITY:
Inclusion Criteria:

* a) English- or Spanish-speaking
* b) maternal age >18 years old
* c) smartphone ownership for remote blood pressure ascertainment
* d) diagnosis of gestational hypertension, preeclampsia, or chronic hypertension at hospital discharge
* e) plan to receive postpartum care at a Women & Infants Hospital (WIH)-affiliated clinic

Exclusion Criteria:

* a) fetal anomaly
* b) prisoners
* c) lack of smartphone
* d) inability to consent.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Anyone who is postpartum--regardless of gender identity--will be eliglble to participate
Enrollment: 120 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lewkowitz, MD, MPHS, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Data from this small pilot will not be made available to other researchers.

REFERENCES:
- [Derived] Lewkowitz AK, Schlichting LE, Ayala NK, O'Neill A, McCleary KD, Hardy EJ, Hamel M, Tuuli MG. Association Between Hispanic Ethnicity and Engagement in a Remote Postpartum Blood Pressure Monitoring Programs: Secondary Analysis of a Pilot Randomized Trial. R I Med J (2013). 2024 Jun 3;107(6):17-18. PMID 38810010

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text-message Based Remote Blood Pressure Monitoring | App-based Remote Blood Pressure Monitoring
Started | 60 | 60
Completed | 60 | 59
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text-message Based Remote Blood Pressure Monitoring | App-based Remote Blood Pressure Monitoring | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 59 | 119
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [28 to 36] | 31 [25 to 34] | 32 [26 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 59 | 119
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 34 | 28 | 62
  Unknown or Not Reported | 17 | 19 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 7 | 18
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 25 | 45
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Ascertainment
Description: Number of participants who adhere to recommended blood pressure check after hospital discharge
Time Frame: 3-10 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Text-message Based Remote Blood Pressure Monitoring | App-based Remote Blood Pressure Monitoring
Number analyzed (Participants) | 60 | 59
Participants | 40 | 39

2. Secondary Outcome: Postpartum Readmission for Hypertension or Preeclampsia
Description: Readmission rate for HTN/preeclampsia
Time Frame: Within 30 days of hospital discharge, patient is readmitted for complications related to hypertension or preeclampsia
Measure: Count of Participants; unit: Participants
Arm/Group | Text-message Based Remote Blood Pressure Monitoring | App-based Remote Blood Pressure Monitoring
Number analyzed (Participants) | 60 | 59
Participants | 4 | 8

3. Secondary Outcome: Adherence to Evidence-based Practice
Description: Medication initiation/titration, postpartum blood pressure goal of <150/100
Time Frame: From randomization until 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Text-message Based Remote Blood Pressure Monitoring | App-based Remote Blood Pressure Monitoring
Number analyzed (Participants) | 60 | 59
Participants | 15 | 16

4. Secondary Outcome: Postpartum Severe Maternal Morbidity Composite
Description: Stroke, seizure/eclampsia, acute fatty liver of pregnancy, posterior reversible encephalopathy syndrome, pulmonary edema, heart failure, hemolysis elevated liver enzymes and low platelets, placental abruption, postpartum hemorrhage, acute kidney injury, transaminitis
Time Frame: From randomization until 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Text-message Based Remote Blood Pressure Monitoring | App-based Remote Blood Pressure Monitoring
Number analyzed (Participants) | 60 | 59
Participants | 0 | 0

5. Secondary Outcome: "Using Any Number From 0 to 10 Where 0 is the Worst Possible Experience and 10 is the Best Possible Experience, Please Rate Your Experience in the Postpartum Hypertension Program"
Description: Patient preference of treatment group
Time Frame: Assessed at randomization and at 40 days postpartum, reported at 40 days postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Text-message Based Remote Blood Pressure Monitoring | App-based Remote Blood Pressure Monitoring
Number analyzed (Participants) | 60 | 59
score on a scale | 10 [9 to 10] | 10 [9 to 10]

6. Secondary Outcome: Decisional Regret Scale
Description: Extent to which participant regrets participating in a treatment group. To help interpret the score more readily with other scales ranging from 0 to 100, these scores can then be converted to a 0-100 scale by subtracting 1 from each item then multiply by 25. To obtain a final score, the items are summed and averaged. A score of 0 means no regret; a score of 100 means high regret.
Time Frame: Assessed at randomization and at 40 days postpartum, reported at 40 days postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Text-message Based Remote Blood Pressure Monitoring | App-based Remote Blood Pressure Monitoring
Number analyzed (Participants) | 60 | 59
score on a scale | 5 [0 to 25] | 0 [0 to 15]

ADVERSE EVENTS:
Time Frame: Adverse data were collected from randomization until study completion (6 weeks postpartum)
Arm/Group | Text-message Based Remote Blood Pressure Monitoring | App-based Remote Blood Pressure Monitoring
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 0/60 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT05595629/Prot_SAP_000.pdf